CLINICAL TRIAL: NCT02763787
Title: A Phase I Study to Investigate the Safety, Tolerability, Pharmacokinetics (Including Food Interaction), and Pharmacodynamics of Single Doses of BIA 3-202 in Healthy Volunteers.
Brief Title: Safety, Tolerability, Pharmacokinetics (Including Food Interaction), and Pharmacodynamics of BIA 3-202
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BIA-3202-01
Record Dates: First submitted 2016-05-04; First posted 2016-05-05 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — nebicapone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (9):
- Placebo (Experimental): Matched placebo was administered in the form of oral tablets, given with 200 ml potable water (single oral doses)
  Interventions: Drug: Placebo
- 10 mg (Experimental): 1 x 10 mg BIA 3-202 tablet BIA 3-202 was administered in the form of oral tablets, given with 200 ml potable water (single oral doses)
  Interventions: Drug: BIA 3-202
- 30 mg (Experimental): 3 x 10 mg BIA 3-202 tablets BIA 3-202 was administered in the form of oral tablets, given with 200 ml potable water (single oral doses)
  Interventions: Drug: BIA 3-202
- 50 mg (Experimental): 5 x 10 mg BIA 3-202 tablets BIA 3-202 was administered in the form of oral tablets, given with 200 ml potable water (single oral doses)
  Interventions: Drug: BIA 3-202
- 100 mg (Experimental): 1 x 100 mg BIA 3-202 tablet BIA 3-202 was administered in the form of oral tablets, given with 200 ml potable water (single oral doses)
  Interventions: Drug: BIA 3-202
- 200 mg (Experimental): 2 x 100 mg BIA 3-202 tablets
  Interventions: Drug: BIA 3-202
- 400 mg (Experimental): 4 x 100 mg BIA 3-202 tablets BIA 3-202 was administered in the form of oral tablets, given with 200 ml potable water (single oral doses)
  Interventions: Drug: BIA 3-202
- 800 mg (Experimental): 8 x 100 mg BIA 3-202 tablets BIA 3-202 was administered in the form of oral tablets, given with 200 ml potable water (single oral doses)
  Interventions: Drug: BIA 3-202
- Food Effect (fed/fasted) (Experimental): 400 mg BIA 3-202: 4 x 100 mg BIA 3-202 tablets BIA 3-202 was administered in the form of oral tablets, given with 200 ml potable water (single oral doses)
  Interventions: Drug: BIA 3-202

INTERVENTIONS:
Drug: BIA 3-202 — single rising oral doses (10 mg, 30 mg, 50 mg, 100 mg, 200 mg, 400 mg, 800 mg)
  Other Names: Nebicapone
  Arms: 10 mg; 100 mg; 200 mg; 30 mg; 400 mg; 50 mg; 800 mg; Food Effect (fed/fasted)
Drug: Placebo — Identical placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of single oral rising doses of BIA 3-202 up to 800 mg (proposed doses 10 mg, 30 mg, 50 mg, 100 mg, 200 mg, 400 mg and 800 mg) in groups of 9 healthy male adult subjects, to characterise the preliminary pharmacokinetics of single rising oral doses of BIA 3-202 in healthy male adult subjects, to investigate the effects of single doses of BIA 3-202 on COMT activity in human erythrocytes and to investigate the effect of food on the pharmacokinetics of a single dose of BIA 3-202.

DETAILED DESCRIPTION:
The study was conducted in two parts, with separate groups of subjects participating in each part.

Part 1 was designed as follows:

* Single centre, Phase I, double-blind, randomised, placebo-controlled study to investigate single rising oral doses of BIA 3-202 of up to 800 mg in sequential groups of nine healthy male adult subjects.
* Within each group of nine subjects, two were to be randomised to receive placebo and the remaining seven were to be randomised to receive BIA 3-202.
* No subject was to be a member of more than one treatment group.
* Doses of BIA 3-202 were to be investigated in ascending order.
* The lowest proposed dose of BIA 3-202 (10 mg) was to be investigated in the first instance.
* Progression to the next higher dose was only to occur if the previous dose level was deemed to be safe and well tolerated by the investigator and the sponsor.
* Following discussion between the investigator and the sponsor an intermediate or repeat dose level could be administered if it was deemed appropriate to increase the safety or scientific value of this first in man exploratory study.
* An appropriate interval of at least 7 days was to separate the investigation of dose levels to permit a timely review and evaluation of safety data prior to proceeding to a higher dose level.

The proposed doses to be used in Part 1 of the study were 10 mg, 30 mg, 50 mg, 100 mg, 200 mg, 400 mg and 800 mg.

In Part 2 of the study, an additional group of eight subjects was to receive a single dose of BIA 3-202, either having fasted overnight or with a high fat meal, in an open label two-way crossover design. Each treatment was to be separated by a period of at least 7 days.

The dose administered in Part 2 was to be determined from the safety and pharmacokinetic data from Part 1 of the study.

Following the review of Part 1 data, protocol amendment 1 was issued, in which it was stated that the dose of BIA 3-202 to be used was 400 mg.

Screening Potential subjects were screened for eligibility within 28 days of admission. Screening consisted of review of medical history, physical examination, neurological examination, vital signs, 12 lead ECG, clinical laboratory safety tests (haematology, coagulation plasma biochemistry, urinalysis, urinary microproteins, HbsAg, anti-HCV and HIV I & II, drugs of abuse and alcohol screen).

Treatment Periods The results of screening were known to the Investigator prior to the subject's admission. On admission the inclusion/exclusion criteria were reviewed and subject written informed consent was obtained.

Eligible subjects were to be admitted to the unit for one treatment period (groups 1-7, in Part 1 of the study) or two treatment periods (group 8, Part 2), on the day prior to receiving trial medication and were to remain in the unit under clinical supervision until at least 24 hours post dose.

BIA 3-202 /placebo was to be administered orally in the morning of day 1.

Safety was to be evaluated by monitoring of adverse events, clinical laboratory safety tests (haematology, biochemistry, coagulation, urinalysis, and urinary microproteins), vital signs, 12-lead ECG, and physical examination, including brief neurological examinations.

Blood samples and urine collections were to be taken at pre-determined time-points for the assay of BIA 3-202 and its metabolite BIA 3-270. Blood samples were also to be taken for the assessment of COMT activity in erythrocytes.

Follow Up Subjects were to attend for a follow up visit 5-7 days following their last discharge. At follow-up, medical history and adverse events were to be reviewed, and clinical laboratory safety tests were to be performed.

ELIGIBILITY:
Inclusion Criteria:

* Adult males aged 18-35 years, with a body mass index (BMI) of 19-28 kg/m2.
* Subjects who were healthy as determined by pre-study medical history, physical examination and 12-lead ECG.
* Subjects who had clinical laboratory tests acceptable to the investigator.
* Subjects who were negative for HbsAg, anti-HCV and HIV I and II tests at screening.
* Subjects who were negative for drugs of abuse and alcohol tests at screening and admission.
* Subjects who were non-smokers for at least 6 months preceding screening.
* Subjects who were able and willing to give written informed consent.

Exclusion Criteria:

* Subjects who did not conform to the above inclusion criteria.
* Subjects who had a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, connective tissue diseases or disorders.
* Subjects who had a clinically relevant surgical history.
* Subjects who had a clinically relevant family history.
* Subjects who had a history of relevant atopy.
* Subjects who had a history of relevant drug hypersensitivity.
* Subjects who had a history of alcoholism.
* Subjects who had a history of drug abuse.
* Subjects who consumed more than 28 units of alcohol a week.
* Subjects who had a significant infection or known inflammatory process on screening and/or admission.
* Subjects who had acute gastrointestinal symptoms at the time of screening and/or admission (e.g. nausea, vomiting, diarrhoea, heartburn).
* Subjects who had an acute infection such as influenza at the time of screening and/or admission.
* Subjects who had used prescription drugs within 4 weeks of first dosing.
* Subjects who had used over the counter medication, excluding routine vitamins but including mega dose vitamin therapy, within one week of first dosing.
* Subjects who had used any investigational drug and/or participated in any clinical trial within 3 months of their first admission to this study.
* Subjects who had previously received BIA 3-202.
* Subjects who had donated and/or received any blood or blood products within 3 months prior to screening.
* Subjects who were vegetarians, vegans and/or had medical dietary restrictions.
* Subjects who could not communicate reliably with the investigator.
* Subjects who were unlikely to co-operate with the requirements of the study.
* Subjects who were unwilling or unable to give written informed consent.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2000-04; Primary Completion 2000-06 (Actual); Study Completion 2000-06

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Pre dose, 15, 30, 60, 90, 120, 150, 180 minutes, 4, 6, 8, 12, 16, and 24 hours post dose.
Time of maximum observed concentration (tmax) | Pre dose, 15, 30, 60, 90, 120, 150, 180 minutes, 4, 6, 8, 12, 16, and 24 hours post dose.
Area under the plasma concentration time curve to last measurable time point (AUC0-t) | Pre dose, 15, 30, 60, 90, 120, 150, 180 minutes, 4, 6, 8, 12, 16, and 24 hours post dose.
Area under the plasma concentration time curve extrapolated to infinity (AUC0-∞) | Pre dose, 15, 30, 60, 90, 120, 150, 180 minutes, 4, 6, 8, 12, 16, and 24 hours post dose.

CONTACTS AND LOCATIONS:
Locations (1):
- Guy's Drug Research Unit (GDRU), London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No